CLINICAL TRIAL: NCT03937076
Title: Efficacy of Intercostal Block Versus Pectoral Nerve Block II in Controlling Acute Post-surgical Pain in Thoracoscopic Surgery
Brief Title: Efficacy of Intercostal Block Versus Pectoral Nerve Block II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Dan Levy Faber, Senior thoracic surgeon, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMC-18-0191-CTIL
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Thoracic Surgical Procedures
Keywords: Intercostal block; Pectoral nerve block II

STUDY DESIGN:
Intervention Model Description: patients will be randomly classified into two groups. In the control group, patients will get intercostal block at the end of the surgery and after then will be treated by the customary postoperative pain control regimen.
  In the research group, patients with get PECS II block at the end of the surgery and will get a similar postoperative pain control regimen.
Who Masked: Participant
Masking Description: Patients will not be informed as to which study group they assigned to. Only the caregivers will have this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intercostal block (No Intervention): patients will get intercostal block at the end of the surgery, control group
- PECS II block (Experimental): patients with get PECS II block at the end of the surgery, research group
  Interventions: Procedure: PECS II block

INTERVENTIONS:
Procedure: PECS II block — Pectoral muscles Nerve block for postsurgical pain, PECS II, based on BUPIVACAINE:
  Pectoral muscles nerve block is a procedure in which local anesthetic is injected into two sites.
  1. between the major and minor pectoral muscles, in order to anesthetize the lateral and medial nerve. This injection is referred to as PECS I block.
  2. between the minor pectoral muscle and the anterior serratus muscle, in order to anesthetize the intercostal nerves.
  Arms: PECS II block

SUMMARY:
The investigators will evaluate the efficacy of two types of pain control blocks in patients going thoracoscopic surgery. Patients will be randomly classified into two groups. In the control group, patients will get intercostal block at the end of the surgery and after then will be treated by the customary postoperative pain control regimen. This group represents the existent treating policy.

In the research group, patients with get PECS II block at the end of the surgery and will get a similar postoperative pain control regimen. The investigators hope to find which pain control block is superior.

DETAILED DESCRIPTION:
Thoracic operations are among the most post-operative painful surgeries. Without a doubt, the emergence of the thoracoscopic approaches has decreased pain severity. The classical methods of pain control that is used in the open thoracic procedures are not suitable in the thoracoscopic milieu. As such, pain control methods should be examined. The most accepted methods are those using different anesthetic blocks based on local anesthetic (Bupivacaine), whether in intercostal block or paravertebral one. Today the investigators use intercostal block consistently in thoracospoic procedures.

Recently, the use of the pectoral nerve block (Pecs II) has emerged for different chest wall surgeries, which has proved to be helpful. As a consequence,the investigators want to examine the efficiency of this block in the control of postoperative pain after thoracoscopic procedures.

In this prospective comparative study, patients will be randomly classified into two groups. In the control group, patients will get intercostal block at the end of the surgery and after then will be treated by the customary postoperative pain control regimen. This group represents the existent treating policy.

In the research group, patients with get PECS II block at the end of the surgery and will get a similar postoperative pain control regimen.

The follow up will include checking the pain level in the postoperative days, the extent of the pain relief medication until the discharge, and patient evaluation at the first post-discharge inspection.

The study will include 40 patients in each arm, which will be older than 18 years without gender limitations. This study will not include people with special demands.

Main inclusion criteria: patients planned for thoracoscopic procedures in the investigators department, capable of understanding, reading and signing on the consent form.

Main exclusion criteria: re-operation in the early post-operative period, re-operation at the same side, a known allergy to BUPIVACAINE.

In the case of conversion from thoracoscopic to open approach, patients will be expelled from the study.

The block will be performed solely by the surgeon or the anesthesiologist. Follow-up period will include the postoperative hospitalization period until the first post-discharge inspection.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for video assisted thoracoscopic surgery
* Over 18 years of age
* No known allergy to Bupivacaine
* Candidate who can read, understand and sign inform consent

Exclusion Criteria:

* Candidate had previous surgery at the same side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
The use of pain medications after surgery | from the end of surgery until participant hospital release, assessed up to 4 weeks
  The amount of pain medications used by each participant in the post surgical period

CONTACTS AND LOCATIONS:
Overall Officials: Dan LEVY FABER, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical center, Haifa, Israel